CLINICAL TRIAL: NCT00873951
Title: Influence of Protein Hydrolysis on Dietary Protein Digestibility and Metabolism in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: Riddet Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Other
Other Study IDs: DEGLAIRE CT
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intact casein (Experimental): Subjects undergo an intestinal and metabolic exploration following the ingestion of a standard mixed meal containing 15% of energy as 15N-labelled intact casein
  Interventions: Other: Intestinal and metabolic exploration; Dietary Supplement: 15N-labelled intact casein
- Hydrolyzed casein (Experimental): Subjects undergo an intestinal and metabolic exploration following the ingestion of a standard mixed meal containing 15% of energy as 15N-labelled hydrolyzed casein
  Interventions: Other: Intestinal and metabolic exploration; Dietary Supplement: 15N-labelled hydrolyzed casein
- AA (Experimental): Subjects undergo an intestinal and metabolic exploration following the ingestion of a standard mixed meal containing 15% of energy as a mixture of AA mimicking the composition of casein but devoid in serine
  Interventions: Other: Intestinal and metabolic exploration; Dietary Supplement: mixture of AA

INTERVENTIONS:
Other: Intestinal and metabolic exploration — Subjects are studied for 8h following the ingestion of a standard meal containing 15% of energy as protein. Intestinal, blood and urine are collected at regular intervals.
Dietary Supplement: 15N-labelled intact casein — standard mixed meal containing 15% of energy as 15N-labelled intact casein
  Arms: Intact casein
Dietary Supplement: 15N-labelled hydrolyzed casein — standard mixed meal containing 15% of energy as 15N-labelled hydrolyzed casein
  Arms: Hydrolyzed casein
Dietary Supplement: mixture of AA — standard mixed meal containing 15% of energy as a mixture of AA mimicking the composition of casein but devoid in serine
  Arms: AA

SUMMARY:
Hydrolysis of dietary protein may impact their gastrointestinal kinetics and further metabolism. The primary goal of this work was to measure the metabolic fate of intact or hydrolyzed protein using a protein of good nutritional quality, i.e., casein. A second aim of this study was to assess the true ileal digestibility of dietary protein using different methods including the hydrolyzed casein method and to measure its possible effect on endogenous intestinal N losses in humans.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects
* BMI between 18 and 25

Exclusion Criteria:

* allergy to dairy proteins
* positive serology to AgHbS, HCV or HIV
* pregnancy
* abusive drug or alcohol consumption.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2006-01; Primary Completion 2006-11 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Postprandial metabolic fate of dietary N | 0h-1h-2h-3h-4h-5h-6h-7h-8h postprandial

SECONDARY OUTCOMES:
Differences in ileal digestibility determination according to the method used | 8h postprandial

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de recherche sur volontaires, Bobigny, France

REFERENCES:
- [Derived] Deglaire A, Moughan PJ, Airinei G, Benamouzig R, Tome D. Intact and hydrolyzed casein lead to similar ileal endogenous protein and amino acid flows in adult humans. Am J Clin Nutr. 2020 Jan 1;111(1):90-97. doi: 10.1093/ajcn/nqz268. PMID 31711108
- [Derived] Deglaire A, Fromentin C, Fouillet H, Airinei G, Gaudichon C, Boutry C, Benamouzig R, Moughan PJ, Tome D, Bos C. Hydrolyzed dietary casein as compared with the intact protein reduces postprandial peripheral, but not whole-body, uptake of nitrogen in humans. Am J Clin Nutr. 2009 Oct;90(4):1011-22. doi: 10.3945/ajcn.2009.27548. Epub 2009 Aug 19. PMID 19692493